CLINICAL TRIAL: NCT01859182
Title: A Multicenter Phase II Study of the Combination of AZD6244 Hydrogen Sulfate and MK-2206 in Patients With Refractory Advanced Biliary Cancers
Brief Title: Selumetinib and Akt Inhibitor MK-2206 in Treating Patients With Refractory or Advanced Gallbladder or Bile Duct Cancer That Cannot Be Removed By Surgery
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-01014; NCI-2013-01014 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OSU 12181 (Other: Ohio State University Medical Center); 9178 (Other: CTEP); N01CM00070 (NIH)
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2013-10

CONDITIONS: Adenocarcinoma of the Gallbladder; Adenocarcinoma With Squamous Metaplasia of the Gallbladder; Adult Primary Cholangiocellular Carcinoma; Advanced Adult Primary Liver Cancer; Cholangiocarcinoma of the Extrahepatic Bile Duct; Localized Unresectable Adult Primary Liver Cancer; Metastatic Extrahepatic Bile Duct Cancer; Recurrent Adult Primary Liver Cancer; Recurrent Extrahepatic Bile Duct Cancer; Stage II Gallbladder Cancer; Stage IIIA Gallbladder Cancer; Stage IIIB Gallbladder Cancer; Stage IVA Gallbladder Cancer; Stage IVB Gallbladder Cancer; Unresectable Extrahepatic Bile Duct Cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Carcinoma, Hepatocellular; Gallbladder Neoplasms | interventions — AZD 6244; MK 2206; Pharmacogenomic Testing

ARMS (1):
- Treatment (selumetinib, Akt inhibitor MK2206) (Experimental): Patients receive Akt inhibitor MK-2206 PO on days 1, 8, 15, and 22 (days 8, 15, and 22 of course 1) and selumetinib PO on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: selumetinib; Drug: Akt inhibitor MK2206; Other: laboratory biomarker analysis; Other: pharmacogenomic studies; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: selumetinib — Given PO
Drug: Akt inhibitor MK2206 — Given PO
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacogenomic studies — Correlative studies
Procedure: quality-of-life assessment — Ancillary studies

SUMMARY:
This phase II trial studies how well selumetinib and Akt inhibitor MK-2206 work in treating patients with refractory or advanced gallbladder or bile duct cancer that cannot be removed by surgery. Selumetinib and Akt inhibitor MK-2206 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the objective response rate (complete response [CR] + partial response [PR]), as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria, in patients with refractory advanced biliary cancers receiving the combination of AZD6244 hydrogen sulfate (selumetinib) and MK-2206 (Akt inhibitor MK-2206).

SECONDARY OBJECTIVES:

I. To determine the overall and progression-free survival in patients with refractory advanced biliary cancer receiving MK-2206 and AZD6244 hydrogen sulfate.

II. To determine the frequency and severity of adverse events and tolerability of AZD6244 hydrogen sulfate + MK-2206 in patients with advanced refractory biliary cancer receiving this regimen.

III. To evaluate the effects of AZD6244 hydrogen sulfate plus MK-2206 on the inflammatory cytokine and immune cell profiles as well as on cancer cachexia.

IV. To determine the presence of genetic mutations of phosphatidylinositol 3 kinase (PI3K)/protein kinase B (Akt) and mitogen-activated protein kinase (MAPK) signaling pathway genes (other than v-raf murine sarcoma viral oncogene homolog [BRAF] V600E) relevant to biliary cancer and how these correlate with and may predict objective response to treatment with AZD6244 hydrogen sulfate and MK-2206.

V. To assess and validate target inhibition in patients with refractory advanced biliary cancer receiving the combination of MK-2206 plus AZD6244 hydrogen sulfate.

VI. To determine the pharmacogenetic profile as a way of assessing inter-individual variability as well as how these relate to clinical outcomes.

VII. To determine genetic variants and mutations in genes encoding drug metabolizing enzymes and transporters, and genes involved in tumor biology, and how these may be related to response to treatment.

VIII. To evaluate the effect of combined MAPK and PI3K/Akt inhibition on skeletal muscle anabolism in patients receiving treatment with AZD6244 hydrogen sulfate and MK-2206.

IX. To conduct quality of life analyses in patients receiving the combination of AZD6244 hydrogen sulfate plus MK-2206.

OUTLINE:

Patients receive Akt inhibitor MK-2206 orally (PO) on days 1, 8, 15, and 22 (days 8, 15, and 22 of course 1) and selumetinib PO on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have surgically unresectable histologically confirmed biliary tract adenocarcinoma (defined as gallbladder cancer, extrahepatic and intrahepatic cholangiocarcinoma; this definition excludes ampullary cancers and all tumors of mixed histology); cytological confirmation is not allowed on this study, as tissue is needed for correlative science; fresh tissue (mandatory) AND paraffin embedded tissue (positron emission tomography [PET]) from tumor blocks (if available) will be required from patients before enrolling on this study
* Patients will be required to undergo a biopsy prior to enrolling on the study and will be given the option to have another biopsy around 4 weeks from initiation of treatment
* Patients must have measurable disease by RECIST 1.1 criteria, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 10 mm with spiral computed tomography (CT) scan (CT scan slice thickness no greater than 5 mm); malignant lymph nodes will be considered measurable if they are >= 15 mm in short axis
* All of the following:

  * Patients must have received only one prior line of systemic therapy for recurrent or advanced disease
  * Prior adjuvant therapy (chemotherapy +/- radiation) completed within 6 months of diagnosis of recurrence/metastases is equivalent to one line of prior therapy for metastatic disease
  * For patients who completed adjuvant therapy > 6 months prior to diagnosis of recurrence/metastases, progression on 1 prior line of systemic therapy for metastatic disease is required
  * No prior Akt inhibitors or mitogen-activated protein kinase kinase (MEK) inhibitors allowed
  * For patients who had having prior cryotherapy, radiofrequency ablation, ethanol injection, transarterial chemoembolization (TACE) or photodynamic therapy, the following criteria must be met

    * 6 weeks must have elapsed since that therapy
    * Indicator lesion(s) is/are outside the area of prior treatment or, if the only indicator lesion is inside the prior treatment area, there must be clear evidence of disease progression associated with that lesion
    * Edges of the indicator lesion are clearly distinct on CT scanning
  * Prior radiation therapy with or without the use of a fluoropyrimidine as a radiosensitizer in the adjuvant setting will be allowed on study if > 12 weeks have elapsed since therapy
  * Prior palliative radiation therapy will be allowed as long as > 2 weeks have elapsed since therapy
* Life expectancy of greater than 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes>= 3,000/µL
* Absolute neutrophil count >= 1,500/µL
* Platelets >= 100,000/µL
* Total bilirubin =< 1.5 X institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal OR =< 5 X institutional upper limit of normal for intrahepatic cholangiocarcinoma if thought to be related to disease
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* The effects of MK-2206 and AZD6244 hydrogen sulfate on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because AZD6244 hydrogen sulfate and MK-2206 is known to be teratogenic, women of childbearing potential and men must use two forms of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, the patient should inform the treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Ability to swallow oral tablets and capsules

Exclusion Criteria:

* Patients who have had chemotherapy, biologic therapy, or immunotherapy, within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events to a grade 1 or less due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-2206 or AZD6244 hydrogen sulfate or other agents used in the study
* Preclinical studies demonstrated the potential of MK-2206 for induction of hyperglycemia in all preclinical species tested; patients with diabetes or in risk for hyperglycemia should not be excluded from trials with MK-2206, but the hyperglycemia should be well controlled on oral agents before the patient enters the trial
* Preclinical studies indicated transient changes in corrected QT (QTc) interval during MK-2206 treatment; prolongation of QTc interval is potentially a safety concern while on MK-2206 therapy; cardiovascular: baseline corrected QT by Fridericia's formula (QTcF) > 450 msec (male) or QTcF > 470 msec (female) will exclude patients from entry on study; a list of medications that may cause QTc interval prolongation should be avoided by patients entering on trial
* Patients with clinically significant bundle branch block or pre-existing clinically significant bradycardia will be excluded from the study
* History of any other malignancy other than biliary cancer in the last 3 years, except for adequately treated basal cell carcinoma, and squamous cell carcinoma of the skin or cervix
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; developmental and reproductive toxicity studies of MK-2206 and AZD6244 hydrogen sulfate have not been performed thus far; women of child-bearing potential and men participating in clinical studies of AZD6244 hydrogen sulfate and MK-2206 must use appropriate contraception, including abstinence and double-barrier methods, throughout AZD6244 hydrogen sulfate and MK-2206 therapy; in preclinical mutagenicity studies, ADZ6244 hydrogen sulfate and MK-2206 were neither genotoxic or mutagenic; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AZD6244 hydrogen sulfate and MK-2206, breastfeeding should be discontinued if the mother is treated with AZD6244 hydrogen sulfate and MK 2206
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with AZD6244 hydrogen sulfate and MK-2206; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Patients requiring strong inhibitors or inducers of cytochrome P450 3A4 (CYP3A4) or those receiving any medications or substances that are inhibitors or inducers of CYP 450 3A4 are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who have a response (PR or CR), assessed by the RECIST v1.1 | 6 months
  Calculated with corresponding 95% binomial confidence intervals.

SECONDARY OUTCOMES:
Frequency and severity of adverse events as per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0 | Up to 4 weeks
  Frequency and severity of adverse events and tolerability of the regimen in each of the patient groups will be collected and summarized by descriptive statistics.
Changes in QOL evaluated using the Functional Assessment of Cancer Therapy - General (FACT-G) | Baseline to 8 weeks
  Changes in overall quality of life will be explored in relation to severe toxicity incidence and in particular to incidence of cachexia. Graphical analyses will be used to assess patterns in these patient reported outcomes in relation to the clinical and tolerability outcomes of incidence.

CONTACTS AND LOCATIONS:
Overall Officials: Tanios Bekaii-Saab, Principal Investigator — Ohio State University